CLINICAL TRIAL: NCT01107470
Title: Age-related Variability of the Efficacy and Tolerability of Alternative Pituitary Suppression Regimens in Follicular Stimulation for Assisted Reproduction Purposes. A Randomised, Prospective, Multi-centre Clinical Trial
Brief Title: Age-related Variability of the Efficacy and Tolerability of Alternative Pituitary Suppression Regimens in ART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); IBSA Institut Biochimique SA (Industry); The Second Hospital of Hebei Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zijiang Chen, Professor, Shandong University
Other Study IDs: chenzj
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2010-04

CONDITIONS: Infertility
Keywords: Infertility IVF ART
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group A1: Age 18-34y (with short protocol)
  Interventions: Drug: hFSH（Fostimon）
- Group A2: age 35-42y ( with short protocol)
  Interventions: Drug: hFSH（Fostimon）
- Group B1: age 18-34y ( with long protocol)
  Interventions: Drug: hFSH（Fostimon）
- Group B2: age 35-42y ( with long protocol)
  Interventions: Drug: hFSH（Fostimon）

INTERVENTIONS:
Drug: hFSH（Fostimon） — After down-regulation (short protocol), all patients will be stimulated with hFSH (human-derived FSH).
  Groups: Group A1
Drug: hFSH（Fostimon） — After down-regulation (short protocol), all patients will be stimulated with hFSH (human-derived FSH).
  Groups: Group A2
Drug: hFSH（Fostimon） — After down-regulation (long protocol), all patients will be stimulated with hFSH (human-derived FSH).
  Groups: Group B1
Drug: hFSH（Fostimon） — After down-regulation (long protocol), all patients will be stimulated with hFSH (human-derived FSH).
  Groups: Group B2

SUMMARY:
Age-related variability of the efficacy and tolerability of alternative pituitary suppression regimens in follicular stimulation for assisted reproduction purposes. A randomised, prospective, multi-centre clinical trial

DETAILED DESCRIPTION:
Pituitary suppression is strongly advised to be included within the follicular stimulation protocols to avoid the occurrence of a premature LH surge, which leads to cycle cancellation.

However, whatever the drug and the schedule selected to achieve it, it is clear that pituitary suppression constitute a major perturbation of the endocrine milieu and that it has an impact on the outcome of the stimulation.

Indeed, the data in the literature support the idea that pituitary down-regulation by GnRH agonists according to the so-called long protocol, resulting in a deeper suppression, result in better clinical outcomes as compared to the short protocol, at least in women of younger reproductive age. Conversely, it has been proposed that a less profound suppression (e.g. short protocol), that allows better background regulation from the pituitary, should be preferred in women of advanced reproductive age.

However, the majority of the data currently supporting the decision makers in selecting their pituitary suppression strategies is based on studies focussed on standard, good prognosis patients whereas just a few studies have specifically addressed the special issue of the advanced reproductive age. Inasmuch, very few data are available in pure (non resistant) advanced age patients and, however, no studies have compared in the same setting younger vs aged subjects with an adequate sample size.

Another intriguing aspect of the question is that the chronological age does not necessarily overlap with the reproductive age which, besides complicating the decisional process in the clinical practise, may also play as a confounding factor in the evaluation of the results from clinical trials. Several studies have validated the role of the so-called follicle antral count (AFC) and the anti-Mullerian hormone (AMH) circulating levels as having a predictive role in the evaluation of the actual reproductive age. In particular the latter, the AMH, appears to be easier to standardise and to be used as the best reference in multicentre clinical studies focussed on the reproductive age.

In summary, there is a clear lack of information on the performance of the different GnRH-agonist schedules in alternative chronological and reproductive age groups and the data from a large size prospective trial may generate valuable indications for the daily clinical practise.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 42
* First IVF attempt
* BMI 18 to 25
* Basal FSH less than 12 for subjects below the age of 35 or less than 15 for subjects aged more than 35
* Informed consent

Exclusion Criteria:

* Genital malformation
* Hypersensitivity to study drugs
* Major illnesses (to be specified)
* PCOS

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients addressed to follicular stimulation for in vitro fertilisation purposes will constitute the study population.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zijiang Chen, Professor, Study Director — Director of Shandong University reproductive medicine study center
Locations (1):
- Shandong University reproductive medicine researche center, Jinan, Shandong, China